CLINICAL TRIAL: NCT04594681
Title: A Phase I Study of KHK4951 in Healthy Volunteers and Patients With Wet Age-Related Macular Degeneration
Brief Title: A Safety Study of KHK4951 in Healthy Volunteers and Patients With Wet Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor judged that the objectives of this Phase 1 study were satisfied, and the study was terminated after the completion of Cohort 3 Step 3.
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4951-001
Record Dates: First submitted 2020-09-22; First posted 2020-10-20 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers; Wet Age-related Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- KHK4951 (Experimental)
  Interventions: Drug: KHK4951

INTERVENTIONS:
Drug: Placebo — Placebo is administered once daily or three times daily.
  Arms: Placebo
Drug: KHK4951 — KHK4951 is administered once daily or three times daily.
  Arms: KHK4951

SUMMARY:
The purpose of this study is to evaluate safety and tolerability after administration of KHK4951 in healthy volunteers and patients with wet age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria: Healthy Volunteers

* Voluntary written informed consent to participate in the study
* Japanese or white men 20 to < 50 years at the time of informed consent
* BMI 18.5 to < 30.0 at screening
* Intraocular pressure (study eye) 10.0 mm Hg to 21.0 mm Hg
* Monocular or binocular visual acuity (corrected visual acuity if correction is required) ≥ 1.0 at screening

Inclusion Criteria: Patients

* Voluntary written informed consent to participate in the study
* Age ≥ 50 years at the time of informed consent
* AMD-associated by active subfoveal CNV lesions in the study eye or juxtafoveal CNV lesions with CNV-associated findings in the fovea in the study eye
* CST ≥ 300 μm in the study eye at screening, as measured by OCT
* BCVA score ≥ 23 letters in the study eye at screening and enrollment, as measured by the ETDRS visual acuity chart
* BCVA score ≥ 58 letters in the non-study eye at screening, as measured by the ETDRS visual acuity chart
* In subjects with prior treatment of the study eye with anti-vascular endothelial growth factor (anti-VEGF) drugs such as Beovu, Eylea, Lucentis, Avastin, or Macugen, presence of response to the anti-VEGF drug(s) as judged by the investigator or subinvestigator based OCT, FA, visual acuity, or other assessment results

Exclusion Criteria: Healthy Volunteers

* Current illness requiring treatment
* History of ophthalmologic laser surgery, ophthalmologic surgery, nasolacrimal duct surgery, orany eyelid surgery affecting flow in the nasolacrimal duct
* History of or current circulatory disease (e.g., cerebrovascular or cardiovascular disease)
* History of or current dry eye
* Abnormal findings on OCT at screening or enrollment examination

Exclusion Criteria: Patients

* Clinical findings or a history of conditions other than wAMD affecting the retina and choroid (e.g., diabetic retinopathy, diabetic macular edema, myopic CNV, retinal vein occlusion, or premacular membrane) in either of the eyes
* Any of the following diseases in the study eye:

  * Glaucoma
  * Ischemic optic neuropathy
  * Retinitis pigmentosa
* Current or history of vitreous hemorrhage or macular hole in the study eye
* Any abnormality in the anterior segment of the eye or vitreous body that may affect fundus observation by OCT, color fundus photography, or fluorescein angiography

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Day 1 to Day 43
  For adverse events that occurred after administration of the investigational drug, number of subjects with AEs and occurrence frequency are evaluated.

SECONDARY OUTCOMES:
Serum KHK4951 concentration | Healthy Volunteers: Day 1, Day2, Day4, Day8, Day12, Day16, Day21, Day23, Day 25, Day 29, Day 36, Day 43; Patients: Day 1, 8, 22, 43
Time to the maximum concentration | Day 1 to Day 43
The maximum concentration | Day 1 to Day 43
Area under the concentration-time curve | Day 1 to Day 43
Apparent clearance | Day 1 to Day 43
Elimination half-life | Day 1 to Day 43

CONTACTS AND LOCATIONS:
Locations (1):
- Hakata clinic, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Undecided